CLINICAL TRIAL: NCT02595593
Title: A Multicenter Prospective Randomized Trial on the Intervention of Rib Fixation for Clinically Severe Rib Fractures From Trauma
Brief Title: Rib Fixation for Clinically Severe Rib Fractures From Trauma
Acronym: SOFRIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Darwin Ang (Other)
Responsible Party: Sponsor-Investigator, Darwin Ang, Director, Medical Trauma Services, Ocala Health Trauma, SCRI Development Innovations, LLC
Organization: SCRI Development Innovations, LLC (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SCRI HEOR_02
Record Dates: First submitted 2015-04-30; First posted 2015-11-03 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Rib Fracture; Flail Chest
Keywords: Trauma; Rib Plate; Rib Fixation
MeSH Terms: conditions — Rib Fractures; Flail Chest; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rib Fixation System (Active Comparator): This group of subjects will receive a surgical rib plating procedure after trauma
  Interventions: Device: Rib Fixation System
- Critical Care and Pain Control (No Intervention): This group will receive critical care and pain control after trauma

INTERVENTIONS:
Device: Rib Fixation System — This intervention involves a surgical procedure to affix rib plates to broken ribs
  Other Names: DePuySynthes MatrixRIB Contoured Rib Implants
  Arms: Rib Fixation System

SUMMARY:
This is a multicenter randomized study investigating the differences in clinical outcomes of patients between two standard of care pathways for rib trauma: patients who receive rib fixation versus patients who receive modern critical care and pain control after sustaining clinically significant rib fractures from trauma.

DETAILED DESCRIPTION:
This study will compare the outcomes of patients between two standard of care pathways for rib trauma: those who have their ribs plated versus those who are managed by modern critical care and pain control. A study nurse (project) coordinator will identify subjects based on inclusion and exclusion criteria, then obtain consent for each of these patients prior to randomization. Randomization will be decided by a web-based computer program, accessible to the project coordinator. Although this randomization occurs, the study itself is purely observational, as the intervention is currently standard of care. None of the subjects or study group members will be blinded since it is not possible to disguise the intervention. Patients will be evaluated and a survey will be administered at set post-intervention intervals to determine endpoints and quality of life when data analysis will also take place.

ELIGIBILITY:
Inclusion Criteria:

* Flail chest, defined as 3 or more consecutive ribs fractured in more than one place
* Pain and disability of an FPS (Functional Pain Scale) rating of 3 or higher
* Deformity and Defect
* Non-Union
* Thoracotomy for other indications
* 3 or more rib fractures with rib displacement of more than 1 rib cortical diameter
* Failure to wean from ventilator

Exclusion Criteria:

* Active bacteremia
* Active shock
* Severe Traumatic Brain Injury with GCS < 8
* Age 17 years or less or age greater than 90 years old
* Chronic pulmonary disease requiring home oxygenation
* Acute Respiratory Distress Syndrome
* Penetrating chest trauma
* Chronic opioid dependence
* Fractures less than 3cm from vertebral spine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
ICU Length of Stay | measured through study completion, up to 2 years
  length of stay in days

SECONDARY OUTCOMES:
Quality of Life, as determined by SF-36 survey | measured at 1 week, 3 months, 6 months post-intervention
  measured at 3 different time points post-hospital stay
Number of participants with pneumonia as defined by the Centers for Disease Control | measured monthly through course of study, up to 2 years
  based on classification as complication of rib trauma treatment
Total cost of treatments | measured through study completion, up to 2 years
  measured based on total costs during length of hospital stay

OTHER OUTCOMES:
Complication Rates | measured at 1 week, 3 months, 6 months
  including, but not limited to, pneumonia, urinary tract infection, arrhythmia, sepsis, reintubation, wound infection
Pain Control documented by the Functional Pain Scale | measured before and after surgery and at time of discharge, through study completion, up to 2 years
  measured using the Functional Pain Scale
Ventilator/Ventilator Free Days | measured through study completion, up to 2 years
  measured in days on or off ventilation, based on length of stay in hospital
Narcotic usage | measured at 1 week, 3 months, 6 months
  converted to units of morphine
Hospital length of stay | measured through study completion, up to 2 years
  measured in days
Pulmonary Function | measured at discharge, 3 months, and 6 months, through study completion, up to 2 years
  as measured by FVC (forced vital capacity), FEV1, and TLC by spirometry
Time to wean from ventilator | measured through study completion, up to 2 years
  measured in days
Tracheostomy rates | measured at 1 week, 3 months, 6 months
  overall rate of tracheostomy in population

CONTACTS AND LOCATIONS:
Overall Officials: Darwin Ang, MD, Principal Investigator — HCA Trauma Network
Locations (10):
- United States (10):
  - Fort Walton Beach Medical Center, Fort Walton Beach, Florida
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Kendall Regional Medical Center, Miami, Florida
  - Ocala Regional Medical Center - Health Trauma, Ocala, Florida
  - Orange Park Medical Center, Orange Park, Florida
  - Central Florida Regional Hospital, Sanford, Florida
  - Research Medical Center, Kansas City, Missouri
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Chippenham Johnston-Willis Hospital, Richmond, Virginia